CLINICAL TRIAL: NCT07320768
Title: The Efficacy and Safety of Renal Denervation Combined With Pulsed Field Ablation in Preventing Blanking Period Recurrence of Atrial Arrhythmia in Patients With Persistent Atrial Fibrillation: An OFF-MED Trial
Brief Title: Renal Denervation Combined With Pulsed Field Ablation to Prevent Blanking-Period Recurrence in Persistent Atrial Fibrillation
Acronym: OFF-MED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Shanghai Shineyo Medical Co., Ltd. (Unknown); BRATTEA Medtech Co. Ltd (Unknown)
Responsible Party: Principal Investigator, Wenzheng Han, Associate Chief Physician; Administrative Deputy Director, Department of Cardiology, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IS25217
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Persistent Atrial Fibrillation; renal denervation (RDN); pulsed-field ablation (PFA)
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pulsed-field ablation alone (Sham Comparator)
  Interventions: Procedure: Pulsed-Field Ablation (PFA)
- renal denervation combined with pulsed-field ablation (Experimental)
  Interventions: Procedure: renal denervation; Procedure: Pulsed-Field Ablation (PFA)

INTERVENTIONS:
Procedure: renal denervation — Renal denervation is a catheter-based procedure performed after renal angiography confirms no significant stenosis. A specialized catheter delivers low-energy pulses inside both renal arteries to disrupt overactive sympathetic nerves surrounding the vessels. Energy is applied in a spiral pattern from distal to proximal segments. The procedure is performed during the same session as PFA under anticoagulation.
  Arms: renal denervation combined with pulsed-field ablation
Procedure: Pulsed-Field Ablation (PFA) — Catheter-based PFA of the left atrium for wide-antral pulmonary vein isolation using a multielectrode PFA system. Entrance/exit block must be confirmed.

SUMMARY:
The goal of this clinical trial is to learn whether adding renal denervation (RDN) to pulsed-field ablation (PFA) reduces blanking-period recurrence of atrial tachyarrhythmias in adults (≥18 years) with persistent atrial fibrillation undergoing first-time ablation while off antiarrhythmic drugs.

The main questions it aims to answer are:

1. Does PFA+RDN, compared with PFA alone, reduce the proportion of participants with any AF/atrial flutter/atrial tachycardia ≥30 seconds during the 90-day blanking period?
2. Is PFA+RDN safe, as measured by procedure-related serious adverse events through 30 days?

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Patients with persistent atrial fibrillation undergoing first-time catheter ablation (defined as any episode lasting ≥7 days).
* Symptomatic atrial fibrillation refractory to or intolerant of at least one class I or III antiarrhythmic drug and scheduled for guideline-directed catheter ablation.
* Able to understand the study purpose, voluntarily participate, and sign the written informed consent form.

Exclusion Criteria:

* Presence of advanced structural heart disease.
* Life expectancy < 12 months.
* Blood pressure < 90/60 mmHg.
* Pregnant or lactating women.
* Anatomical abnormalities of the renal arteries unsuitable for treatment as determined by pre-procedural renal CTA.
* History of renal artery intervention, impaired renal function with estimated glomerular filtration rate (eGFR) < 45 mL/min/1.73 m² (calculated by the MDRD equation).
* Secondary atrial fibrillation due to electrolyte imbalance, thyroid disorders, or other reversible or non-cardiac causes.
* Contraindication to pulsed-field ablation (e.g., left atrial thrombus, prior atrial septal defect occluder implantation, or permanent metallic implant in the left atrium) or to anticoagulation therapy.
* Known inability to obtain vascular access or contraindication to femoral venous puncture.
* Heart failure with left ventricular ejection fraction < 30% documented by transthoracic echocardiography within 3 months before ablation.
* Patients with current or anticipated need for pacemaker, implantable cardioverter-defibrillator (ICD), or cardiac resynchronization therapy (CRT), or prior transseptal closure with occluder device for atrial septal defect or patent foramen ovale.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 86 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from Atrial Arrhythmia Recurrence | within 12 Months After the Index Procedure
  Absence of any documented atrial tachyarrhythmia - including atrial fibrillation (AF), atrial tachycardia (AT), or atrial flutter (AFL) lasting ≥30 seconds - occurring

SECONDARY OUTCOMES:
Freedom from AF recurrence | within 3 months after the index procedure
  Absence of any documented atrial fibrillation (AF) episode lasting ≥ 30 seconds after a single ablation procedure, without use of antiarrhythmic drugs during follow-up.
Atrial fibrillation burden | at 3 months
  AF burden measured by 24-hour (or longer) Holter monitoring at 3 months, calculated as the proportion of AF duration to total recording time, in participants not receiving antiarrhythmic drugs.
Change in blood pressure | immediately, at 1 month, and at 3 months after procedure
  Change in systolic and diastolic blood pressure from baseline to post-procedure, 1-month, and 3-month follow-up visits.
Major adverse cardiovascular events (MACE) | up to 12 months after ablation
  Incidence of death, stroke, heart failure, major bleeding, non-stroke thromboembolic events, and cardiovascular hospitalization, reported both as individual and composite outcomes.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Heradien M, Mahfoud F, Greyling C, Lauder L, van der Bijl P, Hettrick DA, Stilwaney W, Sibeko S, Jansen van Rensburg R, Peterson D, Khwinani B, Goosen A, Saaiman JA, Ukena C, Bohm M, Brink PA. Renal denervation prevents subclinical atrial fibrillation in patients with hypertensive heart disease: Randomized, sham-controlled trial. Heart Rhythm. 2022 Nov;19(11):1765-1773. doi: 10.1016/j.hrthm.2022.06.031. Epub 2022 Jun 30. PMID 35781044
- [Result] Steinberg JS, Shabanov V, Ponomarev D, Losik D, Ivanickiy E, Kropotkin E, Polyakov K, Ptaszynski P, Keweloh B, Yao CJ, Pokushalov EA, Romanov AB. Effect of Renal Denervation and Catheter Ablation vs Catheter Ablation Alone on Atrial Fibrillation Recurrence Among Patients With Paroxysmal Atrial Fibrillation and Hypertension: The ERADICATE-AF Randomized Clinical Trial. JAMA. 2020 Jan 21;323(3):248-255. doi: 10.1001/jama.2019.21187. PMID 31961420
- [Result] Turagam MK, Whang W, Miller MA, Neuzil P, Aryana A, Romanov A, Cuoco FA, Mansour M, Lakkireddy D, Michaud GF, Dukkipati SR, Cammack S, Reddy VY. Renal Sympathetic Denervation as Upstream Therapy During Atrial Fibrillation Ablation: Pilot HFIB Studies and Meta-Analysis. JACC Clin Electrophysiol. 2021 Jan;7(1):109-123. doi: 10.1016/j.jacep.2020.08.013. Epub 2020 Oct 28. PMID 33478702
- [Result] Romanov A, Pokushalov E, Ponomarev D, Strelnikov A, Shabanov V, Losik D, Karaskov A, Steinberg JS. Pulmonary vein isolation with concomitant renal artery denervation is associated with reduction in both arterial blood pressure and atrial fibrillation burden: Data from implantable cardiac monitor. Cardiovasc Ther. 2017 Aug;35(4). doi: 10.1111/1755-5922.12264. PMID 28423234
- [Result] Pokushalov E, Romanov A, Corbucci G, Artyomenko S, Baranova V, Turov A, Shirokova N, Karaskov A, Mittal S, Steinberg JS. A randomized comparison of pulmonary vein isolation with versus without concomitant renal artery denervation in patients with refractory symptomatic atrial fibrillation and resistant hypertension. J Am Coll Cardiol. 2012 Sep 25;60(13):1163-70. doi: 10.1016/j.jacc.2012.05.036. Epub 2012 Sep 5. PMID 22958958
- [Result] Hering D, Lambert EA, Marusic P, Walton AS, Krum H, Lambert GW, Esler MD, Schlaich MP. Substantial reduction in single sympathetic nerve firing after renal denervation in patients with resistant hypertension. Hypertension. 2013 Feb;61(2):457-64. doi: 10.1161/HYPERTENSIONAHA.111.00194. Epub 2012 Nov 19. PMID 23172929
- [Result] Duytschaever M, Demolder A, Phlips T, Sarkozy A, El Haddad M, Taghji P, Knecht S, Tavernier R, Vandekerckhove Y, De Potter T. PulmOnary vein isolation With vs. without continued antiarrhythmic Drug trEatment in subjects with Recurrent Atrial Fibrillation (POWDER AF): results from a multicentre randomized trial. Eur Heart J. 2018 Apr 21;39(16):1429-1437. doi: 10.1093/eurheartj/ehx666. PMID 29211857
- [Result] Kirchhof P, Camm AJ, Goette A, Brandes A, Eckardt L, Elvan A, Fetsch T, van Gelder IC, Haase D, Haegeli LM, Hamann F, Heidbuchel H, Hindricks G, Kautzner J, Kuck KH, Mont L, Ng GA, Rekosz J, Schoen N, Schotten U, Suling A, Taggeselle J, Themistoclakis S, Vettorazzi E, Vardas P, Wegscheider K, Willems S, Crijns HJGM, Breithardt G; EAST-AFNET 4 Trial Investigators. Early Rhythm-Control Therapy in Patients with Atrial Fibrillation. N Engl J Med. 2020 Oct 1;383(14):1305-1316. doi: 10.1056/NEJMoa2019422. Epub 2020 Aug 29. PMID 32865375
- [Result] Piccini JP, Caso V, Connolly SJ, Fox KAA, Oldgren J, Jones WS, Gorog DA, Durdil V, Viethen T, Neumann C, Mundl H, Patel MR; PACIFIC-AF Investigators. Safety of the oral factor XIa inhibitor asundexian compared with apixaban in patients with atrial fibrillation (PACIFIC-AF): a multicentre, randomised, double-blind, double-dummy, dose-finding phase 2 study. Lancet. 2022 Apr 9;399(10333):1383-1390. doi: 10.1016/S0140-6736(22)00456-1. Epub 2022 Apr 3. PMID 35385695
- [Result] Lin HJ, Wolf PA, Kelly-Hayes M, Beiser AS, Kase CS, Benjamin EJ, D'Agostino RB. Stroke severity in atrial fibrillation. The Framingham Study. Stroke. 1996 Oct;27(10):1760-4. doi: 10.1161/01.str.27.10.1760. PMID 8841325
- [Result] Noubiap JJ, Feteh VF, Middeldorp ME, Fitzgerald JL, Thomas G, Kleinig T, Lau DH, Sanders P. A meta-analysis of clinical risk factors for stroke in anticoagulant-naive patients with atrial fibrillation. Europace. 2021 Oct 9;23(10):1528-1538. doi: 10.1093/europace/euab087. PMID 34279604
- [Result] Benjamin EJ, Wolf PA, D'Agostino RB, Silbershatz H, Kannel WB, Levy D. Impact of atrial fibrillation on the risk of death: the Framingham Heart Study. Circulation. 1998 Sep 8;98(10):946-52. doi: 10.1161/01.cir.98.10.946. PMID 9737513
- [Result] Du X, Guo L, Xia S, Du J, Anderson C, Arima H, Huffman M, Yuan Y, Zheng Y, Wu S, Guang X, Zhou X, Lin H, Cheng X, Dong J, Ma C. Atrial fibrillation prevalence, awareness and management in a nationwide survey of adults in China. Heart. 2021 Jan 28;107(7):535-41. doi: 10.1136/heartjnl-2020-317915. Online ahead of print. PMID 33509976
- [Result] Kalman JM, Sanders P, Rosso R, Calkins H. Should We Perform Catheter Ablation for Asymptomatic Atrial Fibrillation? Circulation. 2017 Aug 1;136(5):490-499. doi: 10.1161/CIRCULATIONAHA.116.024926. PMID 28760871
- [Result] Calkins H, Hindricks G, Cappato R, Kim YH, Saad EB, Aguinaga L, Akar JG, Badhwar V, Brugada J, Camm J, Chen PS, Chen SA, Chung MK, Nielsen JC, Curtis AB, Davies DW, Day JD, d'Avila A, de Groot NMSN, Di Biase L, Duytschaever M, Edgerton JR, Ellenbogen KA, Ellinor PT, Ernst S, Fenelon G, Gerstenfeld EP, Haines DE, Haissaguerre M, Helm RH, Hylek E, Jackman WM, Jalife J, Kalman JM, Kautzner J, Kottkamp H, Kuck KH, Kumagai K, Lee R, Lewalter T, Lindsay BD, Macle L, Mansour M, Marchlinski FE, Michaud GF, Nakagawa H, Natale A, Nattel S, Okumura K, Packer D, Pokushalov E, Reynolds MR, Sanders P, Scanavacca M, Schilling R, Tondo C, Tsao HM, Verma A, Wilber DJ, Yamane T. 2017 HRS/EHRA/ECAS/APHRS/SOLAECE expert consensus statement on catheter and surgical ablation of atrial fibrillation. Heart Rhythm. 2017 Oct;14(10):e275-e444. doi: 10.1016/j.hrthm.2017.05.012. Epub 2017 May 12. No abstract available. PMID 28506916